CLINICAL TRIAL: NCT02805855
Title: Safety and Feasibility of Autologous Culture Expanded Adipose Derived Mesenchymal Stromal Cells in the Treatment of Painful Knee Osteoarthritis
Brief Title: Autologous Culture Expanded Mesenchymal Stromal Cells for Knee Osteoarthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jacob L. Sellon, M.D. (Other)
Responsible Party: Sponsor-Investigator, Jacob L. Sellon, M.D., Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-008179
Record Dates: First submitted 2016-06-16; First posted 2016-06-20 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- S50 (Experimental): Subjects in the S50 cohort will receive one injection of 50 million AMSCs.
  Interventions: Drug: Autologous Adipose-Derived Mesenchymal Stromal Cells
- S100 (Experimental): Subjects in the S100 cohort will receive one injection of 100 million AMSCs.
  Interventions: Drug: Autologous Adipose-Derived Mesenchymal Stromal Cells
- M50 (Experimental): Subjects in the M50 cohort will receive three injections of 50 million AMSCs at one-month intervals.
  Interventions: Drug: Autologous Adipose-Derived Mesenchymal Stromal Cells
- M100 (Experimental): Subjects in the M100 cohort will receive three injections of 100 million AMSCs at one-month intervals.
  Interventions: Drug: Autologous Adipose-Derived Mesenchymal Stromal Cells

INTERVENTIONS:
Drug: Autologous Adipose-Derived Mesenchymal Stromal Cells — Human, autologous, culture expanded, adipose derived, mesenchymal stromal cells (AMSCs) produced on site in the Mayo Clinic Human Cellular Therapy Laboratory using current good manufacturing practices (cGMPs).
  Other Names: AMSCs

SUMMARY:
The study seeks to determine the safety and feasibility of using adipose-derived mesenchymal stromal cells to treat symptoms of mild to severe knee osteoarthritis.

DETAILED DESCRIPTION:
Interventions to alter the natural course of osteoarthritis (OA) in the knee are elusive and joint replacement remains the definitive management for refractory, end-stage disease. The Mayo Clinic has a large, ongoing experience using autologous adipose derived mesenchymal stromal cells (AMSCs) for the treatment of a variety of other diseases under INDs. Thus far, the treatments have been well tolerated. These data along with the investigators' pre-clinical animal studies and published experiences using related approaches lead the investigators to believe that this approach provides a reasonable safety profile to treat patients with refractory painful knee OA. The purpose of the current study is to investigate the safety and feasibility of single and multiple injections of autologous, culture expanded AMSCs in subjects with painful, refractory knee OA. Subjects with unilaterally symptomatic mild to severe knee OA will be enrolled based on satisfaction of inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria

1. Male or female ages 40-70 years

   * Females of childbearing potential must have a negative pregnancy test prior to receiving the study drug and will agree use adequate contraception (hormonal or barrier method or abstinence) from the time of screening to a period of 1 year following completion of the drug treatment cycle. Females of childbearing potential are defined as premenopausal and not surgically sterilized, or post-menopausal for fewer than 2 years. A urine pregnancy test will be performed prior to the administration of the study drug to confirm negative results. If the urine pregnancy test is positive, the study drug will not be administered and the result will be confirmed by a serum pregnancy test. Serum pregnancy tests will be performed at a central clinical laboratory, whereas urine pregnancy tests will be performed by qualified personnel using kit
   * Females becoming pregnant during the study will continue to be monitored for the duration of the study or completion of the pregnancy, whichever is longer. Monitoring will include perinatal and neonatal outcome. Any SAEs associated with pregnancy will be recorded. Females in the multiple-dose cohorts (M50 and M100) who become pregnant during the treatment cycle will not receive their remaining injections.
2. Chronic (> 3 months), unilaterally symptomatic, primary femorotibial knee OA
3. Radiographic medial and/or lateral femorotibial knee OA at least Kellgren-Lawrence grade 2 accompanied by definite joint space narrowing as agreed upon by two study co-investigators
4. Previous 6 week or longer trial of one of the following conservative treatments: activity modification, weight loss, physical therapy, anti-inflammatory medications or injection therapy (e.g. cortisone, hyaluronic acid/viscosupplement)
5. Able to routinely walk without assistance (e.g. cane, walker)
6. Clinically stable target knee
7. No surgery planned in the target knee for at least 12 months following the last injection
8. Completed general physical evaluation with primary care provider within 12 months of enrollment
9. Fully understanding of the requirements of the study and willingness to comply with the treatment plan, including fat harvesting, laboratory tests, diagnostic imaging, repeated knee injections/aspirations, arthroscopic examination and follow-up visits and assessments
10. Can provide written informed consent and complete HIPAA documentation after the nature of the study is fully explained and prior to any study-related procedure

Exclusion Criteria

1. Pregnant or nursing, or planning on becoming pregnant during the study period
2. Congenital or acquired malformation of the target knee resulting in significant deformity or leading to problems with the study treatment or analysis of the results
3. Significant malalignment on full length, standing radiographs
4. Arthroplasty hardware or implantable devices in the index knee (intraosseous screws or other hardware not contacting the articular space are not excluded)
5. Surgery on the index knee within 1 year of study enrollment
6. Injections of any into the index knee within 3 months prior to study enrollment
7. Locking, catching, give-away or another major mechanical symptoms of the target knee
8. Symptomatic patellofemoral arthritis or chondromalacia in the index knee
9. History of intra-articular infection in the index knee
10. History of superficial infection in the index knee within 6 months of study enrollment, or evidence of current superficial infection affecting the index knee
11. History of falls requiring medical attention, or gait instability
12. Clinically significant abnormal hematology (complete blood count with differential), blood chemistry, or urinalysis screening laboratory results, including aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), bilirubin, creatinine, and CRP
13. Body mass index (BMI) > 40 kg/m2
14. Taking anticoagulant medications (e.g. warfarin, heparin) or clopidogrel (Plavix)
15. Taking herbal therapies or supplements within 4 weeks of enrollment or unwilling to avoid use of herbal therapies or supplements until at least 30 days following completion of the study drug treatment cycle (includes, but not limited to chondroitin sulfate, diacerein, n-glucosamine, piascledine, and capsaicin)
16. Taking non-steroidal anti-inflammatory medications (e.g. COX-2 inhibitors) without a stable dosing regimen for at least 4 weeks before baseline evaluation, or anticipating not remaining on a stable dose until at least 30 days following completion of the study drug treatment cycle
17. Use of electrotherapy or acupuncture for OA, unless there is a stable regimen for at least 4 weeks before baseline assessment
18. Taking anti-rheumatic disease medication (including methotrexate or other antimetabolites) within 3 months prior to study enrollment
19. On chronic, immunosuppressive transplant therapy or having a chronic, immunosuppressive state, including use of systemic steroids/corticosteroids
20. Current tobacco product use, including nicotine patch or other nicotine products
21. Systemic inflammatory, rheumatological or connective tissue disorder including but not limited to rheumatoid arthritis, systemic sclerosis, system lupus erythematosus, and Ehlers-Danlos Syndrome
22. Rheumatological or inflammatory disease of the knee or chondrocalcinosis/calcium pyrophosphate disease (CPPD), hemochromatosis, inflammatory arthritis, arthropathy of the knee associated with juxta-articular Paget's disease of the femur or tibia, ochronosis, hemophilic arthropathy, infectious arthritis, Charcot's knee joint, villonodular synovitis, and synovial chondromatosis
23. Ongoing infectious disease, including but not limited to tuberculosis, HIV, hepatitis, and syphilis
24. Clinically significant cardiovascular (e.g. history of myocardial infarction, congestive heart failure or uncontrolled hypertension > 90 mmHg diastolic and/or 180 mmHg systolic), neurologic (e.g. stroke, TIA) renal, hepatic, orthopedic (e.g. surgery on other weight bearing joints that will interfere with study, osteoporosis, acute lower body fractures), or endocrine disease (e.g. diabetes).
25. Vascular or neurological disorder affecting the index either lower limb
26. History of cancer/malignancy with the exception of adequately treated basal cell or squamous cell carcinoma of the skin not associated with the target knee
27. History of blood dyscrasia, including but not limited to anemia, thrombocytopenia, and monoclonal gammopathy
28. Participation in a study of an experimental drug or medical device within 3 months of study enrollment
29. Known allergy to local anesthetics of other components of the study drug
30. Any contraindication to MRI scan according to MRI guidelines, or unwillingness to undergo MRI procedures
31. History of or current evidence of alcohol or drug abuse or dependence, recreational use of illicit drug or prescription medications, or have use of medical marijuana within 30 days of study entry
32. Any illness or condition which, in the investigators' judgement will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-10-26 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing adverse events. | 2 years post final injection
  Assess the local and systemic safety of single and multiple injections of human, autologous, culture expanded AMSCs in the treatment of symptomatic knee OA.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Sellon, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials